CLINICAL TRIAL: NCT03273114
Title: Cognitive Functional Therapy (CFT) Compared With a Combined Core Training Exercise and Manual Therapy (CORE-MT) in Patients With Non-specific Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Cognitive Functional Therapy (CFT) Compared With Core Training Exercise and Manual Therapy (CORE-MT) in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Ney Armando Meziat Filho, Assistant Professor, Rehabilitation Sciences, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: neymeziat
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain; Back Pain; Pain; Signs and Symptoms; Neuromuscular Manifestations
Keywords: back pain; physiotherapy; exercise therapy; cognitive functional therapy; low back pain; backache; lower back pain; lumbago; multidimensional; biopsychosocial
MeSH Terms: conditions — Low Back Pain; Back Pain; Pain; Signs and Symptoms; Neuromuscular Manifestations | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with concealed allocation, blinded assessor, blinded participants and intention to treat analysis. Patients will be evaluated at baseline, 8 weeks, 6 and 12 months after randomization, to assess the maintenance of any effect of treatment. The patients in the CFT group will be treated by a physical therapists that attended twice the CFT workshops with two of the tutors of the method. She completed 106 hours of training including workshops, patient examinations and a pilot study with the supervision of a physical therapist with more than three years of clinical experience in CFT. Patients in CORE group will be treated by a physical therapist with clinical experience in manual therapy and core training exercises.
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical outcomes will be obtained in the evaluations carried out by a blinded assessor 8 weeks, 6 and 12 months after randomization. Both arms include active treatments, and participants will not know whether they are in the experimental group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy (CFT) (Experimental): Cognitive Functional Therapy (CFT) is a behavioral intervention that addresses multiple aspects of low back pain. This approach focuses on changing the patient's beliefs, confronting their fears, educating them about pain mechanisms, increasing mental strength, and control of their body. This is done with functional tasks performed by individuals training them to reduce excessive muscle activity in the trunk and generate behavioral changes related to pain, from postures and provocative movements.
  Interventions: Behavioral: Cognitive Functional Therapy
- Core Training Exercise and Manual Therapy (CORE-MT) (Active Comparator): The active comparator will be the combination of Core Training Exercise and Manual Therapy (CORE-MT).
  Interventions: Other: Core Training Exercise and Manual Therapy

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy — There will be four main components in the intervention, following the protocol used by O'Keefe et al. (2015):
  1. The cognitive component will focus on on the multidimensional nature of persistent pain about individual beliefs, and how emotions and behaviors (movement and lifestyle) can reinforce a vicious cycle of pain and disability.
  2. Specific Functional training is designed to normalize maladaptive or provocative movement and posture.
  3. Functional integration directed to activities of daily life that are avoided by the patient (rolling in bed, sitting, sitting to standing, walking, bending and lifting)
  4. Patients will be advised to gradually increase physical activity based on their preference, also focusing on sleep hygiene, stress, and management strategies
  Arms: Cognitive Functional Therapy (CFT)
Other: Core Training Exercise and Manual Therapy — According to the pragmatic clinical decision of the physiotherapist responsible for this intervention arm, participants allocated to the comparison group will be treated with active exercises will involve contractions of abdominal and back muscles in different functional positions, as well as joint mobilization or manipulation techniques applied to the lower back or pélvis, when necessary. Most patients in this group will receive exercises to perform at home, but not related to CFT.
  Arms: Core Training Exercise and Manual Therapy (CORE-MT)

SUMMARY:
There is evidence, of a single randomized controlled trial, that CFT is better than combined manual therapy and motor control exercise for chronic low back pain. However, this study had significant methodological shortcomings regarding the failure to carry out the intention to treat analysis and a considerable loss of follow-up of patients. As it is, it is important to carry out more studies involving CFT compared to other interventions already used in clinical practice and to correct these methodological shortcomings. Therefore, the aim of the study is to assess the efficacy of Cognitive Functional Therapy in patients with chronic non specific low back pain.

DETAILED DESCRIPTION:
Randomized controlled trial with concealed allocation, blinded assessor, blinded participants and intention to treat analysis. Patients will be evaluated at baseline, 8 weeks, 6 and 12 months after randomization, to assess the maintenance of any effect of treatment. The patients in the CFT group will be treated by a physical therapists that attended twice the CFT workshops with two of the tutors of the method. She completed 106 hours of training including workshops, patient examinations and a pilot study with the supervision of a physical therapist with more than three years of clinical experience in CFT. Patients in CORE-MT group will be treated by a physical therapist with clinical experience in manual therapy and core training exercises.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Low back pain for more than 3 months
* Disability score of 14% or more on the Oswestry Disability Index (ODI)
* Being able to walk independently with or without support
* Understand Portuguese well enough to be able to fill in the questionnaires

Exclusion Criteria:

* Main pain area is not the lumbar spine (from T12 to buttocks)
* Main pain as leg pain (eg: nerve root compression or herniated disc with radicular pain / radiculopathy, lateral and central stenosis)
* Less than 6 months after lumbar spine, lower limb or abdomen surgery
* Invasive procedures for pain relief (ex: epidural injection, rhizotomy) in the last 3 months
* Pregnancy
* Inflammatory/rheumatological diseases (e.g., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, systemic lupus erythematosus, Scheuermann's disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  It will be measured by the Brazilian version of the Numerical Scale of Pain 11 points (END). The END scale goes from 0 to 10, where 0 is "no pain" and 10 is "the worst pain imaginable." Participants will be asked to answer about their pain levels based on the last seven days
Disability associated to low back pain | 8 weeks
  It will be assessed by the Brazilian version of the Oswestry Disability Index (ODI). It is a tool widely used in research and clinical practice to assess the disability low back pain. This questionnaire has 10 items (0-5 points each) related to activities of daily living that patients with low back pain have more difficulties to do. The sum of the scores of items is multiplied by two and the percentage of disability varies from 0 to 100 %.

SECONDARY OUTCOMES:
Global impression of recovery | 8 weeks, 6 and 12 months after randomization
  It will be evaluated based on the Global Perceived Effect Scale (GPES) which is an 11-point scale ranging from -5 ('vastly worse'), through 0 (no change) to +5 (completely recovered).
Pain intensity | 6 and 12 months after randomization
  It will be measured by the Brazilian version of the Numerical Scale of Pain 11 points (END) 13. The END scale goes from 0 to 10, where 0 is "no pain" and 10 is "the worst pain imaginable." Participants will be asked to answer about their pain levels based on the last seven days.
Disability associated to low back pain | 6 and 12 months after randomization
  It will be assessed by the Brazilian version of the Oswestry Disability Index (ODI). It is a tool widely used in research and clinical practice to assess the disability low back pain. This questionnaire has 10 items (0-5 points each) related to activities of daily living that patients with low back pain have more difficulties to do. The sum of the scores of items is multiplied by two and the percentage of disability varies from 0 to 100 %.
Patient Satisfaction (mediator of outcome) | 8 weeks, 6 and 12 months after randomization
  This is a simple questionnaire from 1 to 5 asking the patients how satisfied they were with their treatment: 1 = satisfied, 2 = just a little satisfied, 3 = neither satisfied nor dissatisfied, 4 = just a little dissatisfied, 5 = dissatisfied
Catastrophization (mediator of outcome) | 8 weeks, 6 and 12 months after randomization
  It will be evaluated by the question "When I feel pain, it's terrible and I feel it's never going to get any better."with the response options ranging from "Never do that" = 0 to "Always do that" = 10.
Depression (mediator of outcome) | 8 weeks, 6 and 12 months months after randomization
  It will be evaluated by the question "During the past month have you often been bothered by feeling down, depressed or hopeless?" with the response options ranging from "Never" = 0 to "All the time" = 10.
Fear of movement (mediator of outcome) | 8 weeks, 6 and 12 months months after randomization
  It will be assessed by the question "Physical activity might harm my back" and the response options will range from 0 ("completely disagree") to 10 ("completely agree).
Stress (mediator of outcome) | 8 weeks, 6 and 12 months months after randomization
  It will be evaluated by the question "Do you feel stressed? and the response options will range from 0 ("completely disagree") to 10 ("completely agree)
Sleep (mediator of outcome) | 8 weeks, 6 and 12 months months after randomization
  It will be evaluated by the question "Did you have sleep problems last month?" based on Subjective Health Complaints Inventory19. The response options will be "Not at all"=0, "A little"=1, "Some"=2, and "Serious"=3

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto da Coluna, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Meziat Filho N. Changing beliefs for changing movement and pain: Classification-based cognitive functional therapy (CB-CFT) for chronic non-specific low back pain. Man Ther. 2016 Feb;21:303-6. doi: 10.1016/j.math.2015.04.013. Epub 2015 Apr 16. PMID 25920336
- [Background] Meziat Filho N, Mendonca R, Nogueira LA. Lack of confidence in the lower limb: Cognitive Functional Therapy (CFT) for a unilateral loading impairment in chronic non-specific low back pain. Case report. Man Ther. 2016 Sep;25:104-8. doi: 10.1016/j.math.2016.02.007. Epub 2016 Mar 12. PMID 27052627
- [Background] Vibe Fersum K, O'Sullivan P, Skouen JS, Smith A, Kvale A. Efficacy of classification-based cognitive functional therapy in patients with non-specific chronic low back pain: a randomized controlled trial. Eur J Pain. 2013 Jul;17(6):916-28. doi: 10.1002/j.1532-2149.2012.00252.x. Epub 2012 Dec 4. PMID 23208945
- [Background] O'Keeffe M, Purtill H, Kennedy N, O'Sullivan P, Dankaerts W, Tighe A, Allworthy L, Dolan L, Bargary N, O'Sullivan K. Individualised cognitive functional therapy compared with a combined exercise and pain education class for patients with non-specific chronic low back pain: study protocol for a multicentre randomised controlled trial. BMJ Open. 2015 Jun 1;5(6):e007156. doi: 10.1136/bmjopen-2014-007156. PMID 26033941
- [Background] Caneiro JP, Smith A, Rabey M, Moseley GL, O'Sullivan P. Process of Change in Pain-Related Fear: Clinical Insights From a Single Case Report of Persistent Back Pain Managed With Cognitive Functional Therapy. J Orthop Sports Phys Ther. 2017 Sep;47(9):637-651. doi: 10.2519/jospt.2017.7371. Epub 2017 Jul 13. PMID 28704623
- [Background] Bunzli S, McEvoy S, Dankaerts W, O'Sullivan P, O'Sullivan K. Patient Perspectives on Participation in Cognitive Functional Therapy for Chronic Low Back Pain. Phys Ther. 2016 Sep;96(9):1397-407. doi: 10.2522/ptj.20140570. Epub 2016 Mar 24. PMID 27013577
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] O'Sullivan P. It's time for change with the management of non-specific chronic low back pain. Br J Sports Med. 2012 Mar;46(4):224-7. doi: 10.1136/bjsm.2010.081638. Epub 2011 Aug 4. No abstract available. PMID 21821612
- [Background] Goyal M, Haythornthwaite JA. Is It Time to Make Mind-Body Approaches Available for Chronic Low Back Pain? JAMA. 2016 Mar 22-29;315(12):1236-7. doi: 10.1001/jama.2016.2437. No abstract available. PMID 27002443
- [Background] Menke JM. Do manual therapies help low back pain? A comparative effectiveness meta-analysis. Spine (Phila Pa 1976). 2014 Apr 1;39(7):E463-72. doi: 10.1097/BRS.0000000000000230. PMID 24480940
- [Background] Kent P, Mirkhil S, Keating J, Buchbinder R, Manniche C, Albert HB. The concurrent validity of brief screening questions for anxiety, depression, social isolation, catastrophization, and fear of movement in people with low back pain. Clin J Pain. 2014 Jun;30(6):479-89. doi: 10.1097/AJP.0000000000000010. PMID 24281277
- [Background] Paungmali A, Joseph LH, Sitilertpisan P, Pirunsan U, Uthaikhup S. Lumbopelvic Core Stabilization Exercise and Pain Modulation Among Individuals with Chronic Nonspecific Low Back Pain. Pain Pract. 2017 Nov;17(8):1008-1014. doi: 10.1111/papr.12552. Epub 2017 Feb 25. PMID 28042685
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Derived] Castro J, Correia L, Donato BS, Arruda B, Agulhari F, Pellegrini MJ, Belache FTC, de Souza CP, Fernandez J, Nogueira LAC, Reis FJJ, Ferreira AS, Meziat-Filho N. Cognitive functional therapy compared with core exercise and manual therapy in patients with chronic low back pain: randomised controlled trial. Pain. 2022 Dec 1;163(12):2430-2437. doi: 10.1097/j.pain.0000000000002644. Epub 2022 Apr 4. PMID 35384931